#### **CONSENT FORM**



**Title:** Investigating the Influence of Mindfulness-Based Intervention on Teachers' Perceived Stress and Psychological Well-being in Rural Indonesia: A Mixed-Method Approach.

# Investigator with the contact number and organisation:

**Dr. Jamilah Hanum Abdul Khaiyom Principal Investigator**Department of Psychology
International Islamic University Malaysia
hanum@iium.edu.my

Ega Asnatasia Maharani
Co-Investigator
Department of Psychology,
International Islamic University Malaysia
+6281802720004 / ega.am@live.iium.edu.my

#### Introduction

We are doing research about stress and psychological well-being which is increase in this country and in this region. I am going to give you information and invite you to be part of this research. You do not have to decide today whether or not you will participate in the research. Before you decide, you can talk to anyone you feel comfortable with about the research.

This consent form may contain words that you do not understand. Please ask me to stop as we go through the information and I will take time to explain. If you have questions later, you can ask them of me or of another researcher

# **Purpose of the Training**

Stress is a problem that causes variety of effects in both teachers' personal and professional life. This Mindfulness-based training is a four-week series of activities aimed at stress management and increasing teachers' psychological well-being. We would like to know how this training affects your stress perception. We also want to learn about your experiences as Mindfulness-based training participants so that this research can help improve teachers' mental health in the future. You will be accompanied by a certified facilitator for four weeks while you learn the concepts and skills of mindfulness.

# Voluntarily Participation.

Your participation in this study is voluntary. It is up to you to decide whether or not to take part in this study. If you decide to take part in this study, you will be asked to sign a consent form. After you sign the consent form, you are still free to withdraw at any time and without giving a reason. Withdrawing from this study will not affect the relationship you have, if any, with the researcher. If you withdraw from the study before data collection is completed, your data will be returned to you or destroyed.

#### **Procedures**

This research will last for a total of one month. During this period, we will meet you in a training format with a duration of 2-2.5 hours / meeting, once a week. The research location is in the Multipurpose Room Ahmad Dahlan University, Yogyakarta. Before and after the study, you will be asked to fill out a questionnaire as part of data collection.

# **Rights and Obligations**

- 1. You have the right to decide whether or not to participate in this activity. Your decision has no effect on anything.
- 2. In the research process, you will be asked for information through interviews and written information through filling out questionnaires. You have the right to refuse or not to answer if in the process of retrieving information there are questions that cause inconvenience.
- 3. You have the right to withdraw at any time if you find any inconvenience during the training process. However, it would be ideal if you could participate in the training activities from beginning to end so that you receive the most benefits and as expected.
- 4. During the training process, you have the right to ask questions and request clarification if something is unclear.
- 5. You are obliged to maintain the confidentiality of your fellow participants by not sharing anything you hear during the training process to outsiders.
- 6. You are required to attend the entire training series consisting of four meetings and continue to practice independently at home.
- 7. You are prohibited from sharing / duplicating / reproducing the contents of this training material without prior permission from the researcher.

# Benefits

- 1. You get knowledge about mindfulness and stress delivered by professionals.
- 2. You will gain the skills to do mindfulness properly.
- 3. You can observe and feel the benefits of mindfulness on yourself, both psychologically and physically.
- 4. You get the opportunity to share experiences with other participants who are in the same situation as you.
- 5. You get the opportunity to take a break for a moment from your daily routine by doing positive and useful activities.
- 6. You get free training opportunities for 4 meetings.
- 7. You can experience an exclusive psychological mentoring process because it only involves a maximum of 20 participants.

#### Risks

This training does not eliminate the possibility of something unpleasant happening to you. This risk arises as a result of your experience coping with various self-emotions such as sadness, shame, anger, guilt, and so on. Another threat can be uncomfortable physical feelings because some parts of this training demand you to sit in a certain position while learning special breathing techniques. If you are exposed to these risks, we will provide psychological support in the form of private counselling. This help is separate from the training implementation, thus, you are not charged any additional fees.

# **Confidentiality**

All written and verbal information you provide will be kept strictly confidential and used only for research purposes. You could write your initials on the questionnaire, but do not include any confidential personal information. Your response will not be recorded anonymously as part of data processing; however, researchers will ensure confidentiality by:

- 1. Assigning code names/numbers for participants that will be used on all research notes and documents
- 2. Keeping notes, interview transcriptions, and any other identifying participant information in a secure location that only researchers will have access to.

Except in circumstances when investigators are obliged by law to use participant data in reporting special incidents, participant data will be kept entirely confidential. These incidents include, but are not limited to, suicide attempts, self-injury, and acts of violence. If data is exposed for any other reason, you have the right to withdraw all data and information provided and file a complaint or statement of objection to the researcher.

#### **Contact Information**

If you have questions at any time about this study, or you experience adverse effects as the result of participating in this study, you may contact the researcher whose contact information is provided on the first page. If you have questions regarding your rights as a research participant, or if problems arise which you do not feel you can discuss with the Primary Investigator, please contact: (0274) 565515 ext. 3310 / kep@uad.ac.id

#### I hereby acknowledge that

- 1. I voluntarily consent to take part in this research study.
- 2. I have fully discussed and understood the purpose and procedures of this study.
- 3. I have been given enough time to ask any questions that I have about the study, and all my questions have been answered to my satisfaction.
- 4. I may be contacted for further consent, including but not limited to changes in the proposed research.
- 5. I can withdraw from the research at any point of time by informing the Principal Investigator and all my research data obtained prior the consent withdrawal may be retained and used for research.
- 6. I will not have any financial benefits that result from the commercial development of this research.
- 7. I agree / do not agree\* to the photo-taking / audio-recording / video-recording of my participation in the research, for monitoring of treatment integrity and therapist competence. I understand that although my name will be not associated with the photographs/video-recordings used in publication/presentation, I may still be identified.

\*Please delete as appropriate

| Consent to be contacted for future research | |
|---|---|
| Yes, I agree to be contacted for future research that I may | be eligible for. |
| I agree to be contacted via: | |
| Phone | <del></del> |
| Mail | |
| Email | |
| Others | |
| No, I do not agree to be contacted for future research. | |
| | <del></del> |
| Name and Signature (Participant) | Date |